CLINICAL TRIAL: NCT06891391
Title: Comparison of Dynamic Neuromuscular Stabilization Exercises and Deep Cervical Muscle Exercises on Muscle Fat Infiltration in Individuals With Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tokyo Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24072
Record Dates: First submitted 2025-03-14; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Non-specific Neck Pain
Keywords: Dynamic neuromuscular stabilization; Deep neck muscle exercise; Fatty infiltration; Medical resonance imaging; Non-specific neck pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Participants will perform three DNS exercise positions based on their ability: the 3-month prone developmental position, the 6-month developmental position, and the quadruped position. Each position will be done 3-6 repetitions and actively held for 30 to 60 seconds. Participants will perform both exercises at home twice daily, adjusting based on their ability and ensuring they do not experience pain.
  Interventions: Other: Dynamic Neuromuscular Stabilization exercises
- Group B (Active Comparator): Participants will perform two types of exercises: Deep Cervical Flexor Training and Deep Cervical Extensor Training. For flexor training, they will lie on their back with a small towel under the suboccipital region and slowly move their head to the inner range. This will be done in sets of 10 repetitions with a 30-second rest between sets. For extensor training, they will sit upright with their hands folded below the occiput, pushing into extension against their hands and holding the posture as long as possible. This exercise consists of 3 sets of 6 repetitions, with a 6-second rest between repetitions and a 30-seconds break between sets. Participants will perform both exercises at home twice in 6 days a week, adjusting based on their ability and ensuring they do not experience pain.
  Interventions: Other: Deep Cervical Muscle exercises

INTERVENTIONS:
Other: Dynamic Neuromuscular Stabilization exercises — DNS is a method used to enhance muscle stability. It is a manual and rehabilitative approach based on developmental kinesiology to optimize the movement system. These exercises optimize internal muscle forces on each spinal segment.
  Arms: Group A
Other: Deep Cervical Muscle exercises — Deep cervical muscle exercises are isometric exercises that strengthen weak muscles without causing discomfort to pain-sensitive structures like ligaments, tendons, or neck joints. This involves contracting specific muscles without changing muscle length or impeding joint movement.
  Arms: Group B

SUMMARY:
This clinical trial study aims to compare the effects of DNS (Dynamic Neuromuscular Stabilization) exercises and deep cervical muscle exercises on fat infiltration, disability, and posture in individuals with chronic non-specific neck pain. The clinical questions of this study are as follows:

* Can DNS and deep cervical muscle exercises decrease muscle fat infiltration?
* Can DNS and deep cervical muscle exercises improve neck disability?
* Can DNS and deep cervical muscle exercises improve neck posture?

Researchers will compare DNS and deep cervical muscle exercises to people with non-specific neck pain. DNS exercises are hypothesized to significantly reduce fat infiltration and improve neck disability and neck posture compared to deep cervical muscle exercises.

The participants will undergo an MRI scan and clinical assessment, such as NDI (Neck Disability Index) and posture checking, before being randomly divided into two groups. The first group will perform DNS exercises, and the second group will engage in deep cervical muscle exercises. Both sets of exercises will be performed for 16 weeks as part of a daily routine. After the 16-week exercises, the participants will undergo a follow-up MRI, NDI, and posture checking.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific neck pain condition for three months or more
* Mild to moderate disability ( more than 10% of NDI)
* Mild to moderate pain level(2-8/10 of NRS)

Exclusion Criteria:

* A history of spine surgery or cervical injury
* Participated in a neck exercise program in the past three months
* Upper extremity problems
* Radiating pain, numbness, and weakness of the upper extremities
* A detectable pathological spinal condition
* Metabolic disorders, diabetes, and hypertension Obesity

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2025-08-29 (Estimated); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
Change of muscle fat infiltration in the flexor and extensor muscles | 16 weeks
  All participants will be conducted a standard MRI of the cervical spine. They will be asked to lie on their backs and maintain a neutral cervical spine position without rotation, lateral flexion, or exaggerated lordosis. A neck coil will be used during the examination to enhance imaging accuracy. MRI will be performed using the SIGNA Premier 3.OT (GE Healthcare Japan) (Repetition time, 8000 ms; Excitation time, 102 ms; Voxel size, 0.4 x 0.4 mm; Field of view, 200 x 200 mm; Thickness, 3.5 mm). Specific neck muscles (Longus Colli + capitis, Multifidus, Semispinalis cervicis, Semispinalis capitis, and Splenius capitis + cervicis) will be mapped and analyzed for fatty infiltration using Miele-lxiv image processing software. The total fatty infiltration for bilateral muscles at different levels in the neck will be calculated.
Change of disability level | 16 weeks
  The Neck Disability Index (NDI) is a 10-question survey that measures how neck pain affects daily life. The patient rates their pain intensity, headaches, and difficulty with personal care, lifting, reading, concentration, work, driving, sleeping, and recreation. A change of 5%-10% is considered meaningful.
Change of posture | 16 weeks
  Shisei-Karte is a Japanese AI-based website that analyzes posture using images. It assesses head posture, including forward and backward tilts and misalignment. The goal is to detect issues like forward head posture. The process has three steps: (1) participants register with basic details, (2) a side-view photo is taken, and (3) the AI analyzes and displays results in about 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Hardianty A.M Abduh, M. Sc, Study Chair — Tokyo Metropolitan University
Locations (1):
- Tokyo Metropolitan University, Arakawa City, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No